CLINICAL TRIAL: NCT03451149
Title: Single-Arm, Single-Center, Pilot Study To Evaluate The Feasibility And Safety Of Transjugular Intrahepatic Portosystemic Shunt (TIPS) Creation For Portal Hypertension Using A Radiofrequency Guidewire With Intravascular Ultrasound Guidance
Brief Title: Feasibility And Safety Of Transjugular Intrahepatic Portosystemic Shunt (TIPS) Creation Using A Radiofrequency Guidewire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Baylis Medical Company (Industry)
Responsible Party: Principal Investigator, Khashayar Farsad, Associate Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: OHSU eIRB # 16296
Record Dates: First submitted 2018-02-16; First posted 2018-03-01 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Portal Hypertension
Keywords: TIPS
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Intervention Model Description: A single group of up to 10 participants will be enrolled to evaluate a radiofrequency wire for cutting through liver parenchyma instead of the standard trocar needle during transjugular intrahepatic portosystemic shunt creation. This will be to test this device for feasibility and not health outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Experimental): Undergo transjugular intrahepatic portosystemic shunt creation using a radiofrequency wire (Powerwire) in lieu of a trocar needle to cut through liver parenchyma
  Interventions: Device: Radiofrequency wire (Powerwire)

INTERVENTIONS:
Device: Radiofrequency wire (Powerwire) — Using a radiofrequency wire in lieu of a needle for penetrating the liver during transjugular intrahepatic portosystemic shunt creation.

SUMMARY:
A novel radiofrequency (RF) wire created by Baylis Medical (Montreal, CAN) is an FDA cleared device commonly used for percutaneous recanalization procedures. This wire has an active tip that delivers focused RF energy and has been applied for many procedures such as percutaneous transseptal left heart access, recanalization of central vein occlusion, recanalization of arterial occlusion, and recanalization of bile duct occlusion. There has been no study investigating the use of the RF wire for TIPS creation in clinical practice with humans. Having promising results of an experimental feasibility investigation in swine, the investigators are seeking to assess the feasibility and safety of the RF wire to cut through tissue in the liver while creating TIPS in the clinical setting.

DETAILED DESCRIPTION:
The transjugular intrahepatic portosystemic shunt procedure (TIPS), first described in 1969 by Rösch et al., has been widely used to treat the complications of portal hypertension such as recurrent variceal hemorrhage and refractory ascites.

In the TIPS procedure, an intrahepatic connection between a hepatic vein and a portal vein branch is created in order to reduce the portal venous pressure. A dedicated device developed for the TIPS procedure, the Rösch-Uchida Transjugular Liver Access Set (RUPS), is widely used for this procedure. The most challenging and time-consuming part of TIPS creation is puncturing the portal vein from the hepatic vein with a long needle trocar. Occasionally in cirrhotic livers, the trocar needle can deflect and not easily pass through the parenchyma. Needle deflection may lead to additional needle passes and potentially increase risk of inadvertent injury to the liver or extracapsular puncture. There is need, therefore, for a device that can easily penetrate dense liver tissue without creating significant trauma.

A novel radiofrequency (RF) wire created by Baylis Medical (Montreal, CAN) is an FDA cleared device commonly used for percutaneous recanalization procedures. This wire has an active tip that delivers focused RF energy and has been applied for many procedures such as percutaneous transseptal left heart access, recanalization of central vein occlusion, recanalization of arterial occlusion, and recanalization of bile duct occlusion.

The investigators have assessed the application of the RF wire for TIPS creation in a swine model. The investigators found that the use of this wire to cut through tissue during TIPS creation is feasible in swine with some potential advantages compared with the current available tools. The RF wire device was well visualized under intravascular ultrasound (IVUS) guidance and could penetrate through the liver parenchyma smoothly and safely. In addition, the RF wire was able to subsequently be used as a working wire to complete the procedure. Advantages in clinical practice with cirrhotic livers would be the relative ease of penetration into a hardened liver compared to the trocar needle, and the additional benefit of being able to use the device as a working wire to minimize the risk of catheter displacement and decrease procedure time.

There has been no study investigating the use of the RF wire for TIPS creation in clinical practice with humans. Having the promising results of the experimental investigation in swine, the investigators are seeking to assess the feasibility and safety of the RF wire to cut through tissue in the liver while creating TIPS in the clinical setting. It is anticipated that the proposed experimental technique using the RF wire would be at least as safe as the current standard technique. The wire diameter, 0.035 inches, is smaller than the traditionally used 0.038 inch needle trocar, and the deposition of RF energy is limited to the wire tip with minimal collateral damage. Risks of complications, such as puncturing unintended structures including the liver capsule, hepatic artery, gallbladder and biliary tree are anticipated to be at least as low as for the standard technique, estimated at about 3-4%. Moreover, these risks may be reduced even further in the experimental technique owing to the use of intravascular ultrasound guidance, enabling direct visualization of the puncture compared to the standard technique using landmarks and reference images under x-ray fluoroscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cirrhosis and portal hypertension meeting at least one indication for elective TIPS creation including refractory ascites, acute variceal bleeding not responsive to endoscopic treatment, prevention of recurrent variceal bleeding, portal hypertensive gastropathy, hepatorenal syndrome, Budd-Chiari syndrome, hepatic hydrothorax, hepatic veno-occlusive disease, and hepatopulmonary syndrome.
2. Patients who agree to undergo TIPS procedure and participate in this clinical study.
3. Age over 20 years

Exclusion Criteria:

1. Patients with a contraindication for TIPS including congestive heart failure, severe tricuspid regurgitation, severe pulmonary hypertension, uncontrolled systemic infection or sepsis and unrelieved biliary obstruction.
2. Patients in whom intravascular ultrasound cannot be used because of venous occlusion.
3. Decisionally impaired patients
4. Need for emergent TIPS creation

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
Feasibility to use the device as anticipated | within 24 hours
  Ability of the device to perform as anticipated
Incidence of device-related adverse events (Safety) | within 24 hours
  No device-related adverse events

SECONDARY OUTCOMES:
Penetrating ability | within 24 hours
  To assess the capability of the RF wire to cut through tissue without significant deflection through parenchyma
Device use as a standard working wire | within 24 hours
  To assess the capability of the RF wire to act as the working wire for delivery of the TIPS set into the portal vein after access.

CONTACTS AND LOCATIONS:
Overall Officials: Khashayar Farsad, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
HIPAA compliant, IRB-approved, non-identifiable information may be provided for research outcomes purposes.
Time Frame: Anytime after study completion, per approved IRB protocol
Access Criteria: IRB-approved protocols for access to data only